CLINICAL TRIAL: NCT05690568
Title: Changes in Functional Movement Scores Associated With Multimodal Chiropractic Care: a Pilot Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland University Kansas City (Other)
Responsible Party: Principal Investigator, Mark Pfefer, Director of Research, Cleveland University Kansas City
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12062021
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Chiropractic

STUDY DESIGN:
Intervention Model Description: single group pilot study to determine feasibility and potential effect size
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-intervention and post-intervention FMS scores (Other): multimodal chiropractic care with FMS scores assessed pre- and post-intervention
  Interventions: Other: multimodal chiropractic care

INTERVENTIONS:
Other: multimodal chiropractic care — functional movement score followed by intervention of multimodal chiropractic care including spinal/extremity manipulation and exercise recommendation

SUMMARY:
Emergency medical services (EMS) personnel are at high risk of injuries, often related to overexertion while lifting or carrying patients or equipment. They require a high level of functional fitness to operate safely and avoid injuries. The purpose of this pilot study was to explore feasibility and assess effects of multimodal chiropractic care on Functional Movement Screen (FMS) scores among EMS students.

DETAILED DESCRIPTION:
EMS students at a local community college voluntarily completed baseline FMS testing. Those who obtained 14 or less, a sign of movement dysfunction, were recruited to participate in a study to evaluate effects of multimodal chiropractic care on FMS scores. Participants received multimodal chiropractic care with an emphasis on spinal manipulation and corrective exercise for up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* current healthy paramedic students;

Exclusion Criteria:

-

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Functional movement screen score (FMS) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pfefer, RN, MS, DC, Principal Investigator — Cleveland University Kansas City
Locations (1):
- Cleveland University Kansas City Chiropractic Health Center, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided